CLINICAL TRIAL: NCT04597879
Title: Study of the Impact of Severe Brain Injury on the Neuro-vascular and Endothelial Regulation of Peripheral Microcirculation.
Brief Title: Impact of Severe Brain Injury on Neuro-vascular and Endothelial Regulation of Peripheral Microcirculation.
Acronym: MicroTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00183-36; 38RC20.014 (Other: Promotor)
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Severe Traumatic Brain Injury; Trauma
Keywords: Brain trauma; Severe traumatic brain injury; Microcirculation; Speckle; Post-occlusive reactive hyperaemia
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe traumatic brain injury
- Severe trauma without brain trauma
- Healthy controls

SUMMARY:
Severe brain injury (SBI) is one of the world's leading causes of death and disability in young adults, but its peripheral vascular consequences in humans are poorly understood.

This prospective, monocentric, pathophysiological study aims to investigate differences in vasoreactivity in the anterior aspect of the contralateral forearm at the most injured cerebral hemisphere between patients with severe head trauma and patients with severe trauma without associated brain injury matched on sex and age (+/- 5 years).

DETAILED DESCRIPTION:
Severe brain injury (SBI) is one of the world's leading causes of death and disability in young adults.

Its impact on cerebral vascularization is well known. At the systemic level, it induces transient dysfunctions that can develop into severe failures, even in cases of isolated SBI. Studies on a mouse model of SBI show alterations in peripheral vascular reactivity that persist over time and are linked to endothelial dysfunction, the mechanism of which is a decoupling of endothelial NO synthase in a context of systemic inflammation. However, no data are available regarding the peripheral vascular consequences of SBI in humans.

The main objective of this prospective, monocentric, pathophysiological study is to determine whether the postocclusive hyperaemic response at the anterior surface of the contralateral forearm to the most injured cerebral hemisphere differs between patients with severe brain injury and patients with severe trauma without associated head injury matched on sex and age (+/- 5 years), by studying the amplitude of post-occlusive hyperaemia (maximum amplitude expressed as percentage of vasodilatation and area under the curve : AUC) as a function of the group.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers :

* Men and women, over 18 years of age
* Affiliation to a social security scheme
* Signed Consent

Patients with Severe Brain Injury :

* Male and female, over 18 years of age
* Isolated severe brain injury, defined by an initial Glasgow score less than or equal to 8.
* Affiliation to a social security scheme
* Signed informed consent

Severe traumatized patients without associated severe brain injury:

* men and women, over 18 years of age
* severe trauma, defined by an Injury Severity Score (ISS) ≥ 16.
* absence of associated severe brain injury, defined by an initial Glasgow score less than or equal to 8.
* affiliation to or beneficiary of a social security scheme
* signed informed consent

Exclusion Criteria:

* Hypersensitivity to lidocaine and/or prilocaine or to amide type local anesthetics or to any of the excipients of the cream.
* History of axillary lymph node dissection, trauma or axillary surgery
* Prohibited treatments and procedures :

  * In patients with head trauma: ongoing treatment with systemic vasodilators (calcium channel blocker, milrinone).
  * In healthy volunteers: no treatment will be authorized other than paracetamol, hormone supplementation (contraceptive pill, hormone therapy, thyroid hormones).
* Pregnant, parturient or breastfeeding women
* Subject in a period of exclusion from another study,
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure,
* Subject having exceeded the annual compensation threshold for testing
* Subject cannot be contacted in case of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients admitted for severe head trauma or severe trauma without associated severe head trauma in intensive care at Grenoble University Hospital.
  * Healthy volunteers recruited through classified ads
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Post-occlusive hyperaemia | 0-60 days
  Maximum amplitude expressed as percentage of vasodilation and area under the curve: AUC

SECONDARY OUTCOMES:
Post-occlusive hyperaemia with local anesthesia | 0-60 days
  Maximum amplitude expressed as percentage of vasodilation and area under the curve: AUC
Current-Induced Hyperaemia | 0-60 days
  Area under the curve expressed as a percentage of the baseline.
Current-Induced Hyperaemia with local anesthesia | 0-60 days
  Area under the curve expressed as a percentage of the baseline.
Local thermal hyperaemia | 0-60 days
  Maximum amplitude of the initial peak expressed as a percentage of the baseline and area under the curve of the delayed plateau.
Local thermal hyperaemia with local anesthesia | 0-60 days
  Maximum amplitude of the initial peak expressed as a percentage of the baseline and area under the curve of the delayed plateau.
Flow amplitude after local cooling | 0-60 days
  Amplitude of initial vasoconstriction averaged over 1 min around the lowest flow value during the first 5 minutes.
Transient venous post-compression hyperaemia | 0-60 days
  Area under the curve and percentage change from baseline.
Study of vasoreactivity in patients with severe brain injury | 0-60 days
  Extent of post-occlusive hyperaemia, current-induced hyperaemia, thermal hyperaemia and cold response in patients with severe brain injury.
Study of vasoreactivity in healthy subjects | Study visit
  Description of the magnitude of post-occlusive hyperaemia, current-induced hyperaemia, thermal hyperaemia and cold response in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Cracowksi, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France